CLINICAL TRIAL: NCT04310332
Title: 1L- vs. 4L-Polyethylene Glycol for Bowel Preparation Before Colonoscopy Among Inpatients: a Propensity Score-matching Analysis.
Brief Title: 1L- vs. 4L-PEG for Bowel Preparation Among Inpatients.
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Lorenzo Fuccio, Professor of Gastroenterology, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: QIPS propensity score matching
Record Dates: First submitted 2020-03-12; First posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Colonoscopy; Hospitalized Patients; Bowel Preparation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1L-PEG: Hospitalized patients who are prescribed colonoscopy with 1L-polyethylene glycole (PEG) plus ascorbic acid as bowel preparation.
  Interventions: Drug: 1L-PEG
- 4L-PEG: Hospitalized patients who are prescribed colonoscopy with 4L-polyethylene glycole (PEG) as bowel preparation.
  Interventions: Drug: 4L-PEG

INTERVENTIONS:
Drug: 1L-PEG — The drug is 1L-PEG plus ascorbic acid (Plenvu®). It will be administered either the day before colonoscopy, or half the day before and half the day of colonoscopy, or the day of colonoscopy.
  Patients are prescribed bowel prep according to local clinical practice and then all undergo colonoscopy. No standardized intervention on bowel prep is applied, as the design of the study is observational.
  Groups: 1L-PEG
Drug: 4L-PEG — The drug is 4L-PEG. It will be administered either the day before colonoscopy, or half the day before and half the day of colonoscopy, or the day of colonoscopy.
  Patients are prescribed bowel prep according to local clinical practice and then all undergo colonoscopy. No standardized intervention on bowel prep is applied, as the design of the study is observational.
  Groups: 4L-PEG

SUMMARY:
Background and aims: Inpatients are at high risk for inadequate colon cleansing. Experts recommend 4L-polyethylene-glycol (PEG) solution because of its effectiveness and safety profile. A higher colon cleansing adequacy rate for a hyperosmolar 1L-PEG plus ascorbate prep has been recently reported in an observational study among more than 1,000 inpatients. Thus, the present study is aimed at determining whether 1L-PEG outperforms 4L-PEG among inpatients, through a propensity score-matching between the two groups in order to correct for confounders.

ELIGIBILITY:
Inclusion Criteria:

* Adult inpatients scheduled for colonoscopy for any indication within the normal process of care.

Exclusion Criteria:

* patients who underwent emergency or elective therapeutic colonoscopies (e.g. polypectomy, endoscopic mucosal resection, endoscopic submucosal dissection)
* patients who underwent bowel preparation outside the hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients who are scheduled a colonoscopy as inpatients.
Sampling Method: Probability Sample
Enrollment: 1004 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Overall colon cleansing efficacy | Outcome will be assessed during colonoscopy
  Proportion of patients with adequate colon cleansing (Boston Bowel Preparation Score ≥2 for each colon segment)
Right colon cleansing efficacy | Outcome is assessed during colonoscopy
  Proportion of patients with adequate colon cleansing in the right colon (Boston Bowel Preparation Score ≥2 in the right colon)

SECONDARY OUTCOMES:
Safety (serum sodium imbalance) | within 12 hours before starting bowel prep intake; the morning of the day after the colonoscopy
  Degree of serum sodium shift (mmol/L) before and after bowel preparation
Safety (serum potassium imbalance) | within 12 hours before starting bowel prep intake; the morning of the day after the colonoscopy
  Degree of serum potassium shift (mmol/L) before and after bowel preparation
Safety (serum calcium imbalance) | within 12 hours before starting bowel prep intake; the morning of the day after the colonoscopy
  Degree of serum calcium shift (mg/dL) before and after bowel preparation
Safety (serum magnesium imbalance) | within 12 hours before starting bowel prep intake; the morning of the day after the colonoscopy
  Degree of serum magnesium shift (mg/dL) before and after bowel preparation
Safety (serum creatinine imbalance) | within 12 hours before starting bowel prep intake; the morning of the day after the colonoscopy
  Degree of serum creatinine shift (mg/dL) before and after bowel preparation
Safety (glomerular filtration rate change) | within 12 hours before starting bowel prep intake; the morning of the day after the colonoscopy
  Degree of change in glomerular filtration rate (mL/min/1.73 m2), before and after bowel preparation
Safety (hematocrit change) | within 12 hours before starting bowel prep intake; the morning of the day after the colonoscopy
  Degree of change in hematocrit (%), before and after bowel preparation

CONTACTS AND LOCATIONS:
Locations (10):
- Italy (10):
  - Policlinico Sant'Orsola-Malpighi, Bologna
  - Digestive Endoscopy Unit, Fondazione Poliambulanza, Brescia
  - UOSD Gastroenterologia ed Endoscopia Digestiva, Azienda USL di Modena, Carpi
  - Gastroenterology Unit, Valduce Hospital, Como
  - Unit of Gastroenterology and Digestive Endoscopy, Forli-Cesena Hospital, AUSL Romagna, Forlì
  - Digestive Endoscopy Unit, Centro Traumatologico-Ortopedico Hospital, Iglesias
  - Department of Gastroenterology, ASST Rhodense, Rho and Garbagnate Milanese Hospital, Milan
  - Gastroenterology and Digestive Endoscopy Unit, Ospedale Maggiore della Carità, Novara
  - Department of Internal Medicine, Gastroenterology and Hepatology Unit, "Guglielmo da Saliceto" Hospital, Piacenza
  - Gastroenterology Unit, S. Maria delle Croci Hospital, Ravenna

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Frazzoni L, Spada C, Radaelli F, Mussetto A, Laterza L, La Marca M, Piccirelli S, Cortellini F, Rondonotti E, Paci V, Bazzoli F, Fabbri C, Manno M, Aragona G, Manes G, Occhipinti P, Cadoni S, Zagari RM, Hassan C, Fuccio L. 1L- vs. 4L-Polyethylene glycol for bowel preparation before colonoscopy among inpatients: A propensity score-matching analysis. Dig Liver Dis. 2020 Dec;52(12):1486-1493. doi: 10.1016/j.dld.2020.10.006. Epub 2020 Oct 21. PMID 33250131